CLINICAL TRIAL: NCT06912932
Title: The Effects of The Exercise Intensity and Rest Duration on Physiological and Perceptual Responses During 4-Second Sprint Interval Exercise
Brief Title: Physiological and Perceptual Responses During 4-Second Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00004240-CR01
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Fitness
Keywords: exercise; cardiovascular fitness; sprint; vo2max; interval training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- 50% Pmax and 15-s rest duration (Active Comparator): Participants used 50% Pmax and 15-s rest duration during 30 bouts of 4-s sprint interval training.
  Interventions: Behavioral: Preventive
- 50% Pmax and 30-s rest duration (Active Comparator): Participants used 50% Pmax and 30-s rest duration during 30 bouts of 4-s sprint interval training.
  Interventions: Behavioral: Preventive
- 50% Pmax and 45-s rest duration4 (Active Comparator): Participants used 50% Pmax and 45-s rest duration during 30 bouts of 4-s sprint interval training.
  Interventions: Behavioral: Preventive
- 75% Pmax and 15-s rest duration (Active Comparator): Participants used 75% Pmax and 15-s rest duration during 30 bouts of 4-s sprint interval training.
  Interventions: Behavioral: Preventive
- 75% Pmax and 30-s rest duration (Active Comparator): Participants used 75% Pmax and 30-s rest duration during 30 bouts of 4-s sprint interval training.
  Interventions: Behavioral: Preventive
- 75% Pmax and 45-s rest duration (Active Comparator): Participants used 75% Pmax and 45-s rest duration during 30 bouts of 4-s sprint interval training.
  Interventions: Behavioral: Preventive
- All-out Pmax and 15-s rest duration (Experimental): Participants used all-out Pmax and 15-s rest duration during 30 bouts of 4-s sprint interval training.
  Interventions: Behavioral: Preventive
- all-out Pmax and 30-s rest duration (Experimental): Participants used all-out Pmax and 30-s rest duration during 30 bouts of 4-s sprint interval training.
  Interventions: Behavioral: Preventive
- all-out Pmax and 45-s rest duration (Experimental): Participants used all-out Pmax and 45-s rest duration during 30 bouts of 4-s sprint interval training.
  Interventions: Behavioral: Preventive

INTERVENTIONS:
Behavioral: Preventive — systematically investigate the acute physiological responses induced by three levels of %Pmax intensities (50% and 75% of Pmax and all-out efforts) with three varying rest periods (15, 30, and 45-s) between thirty 4-s sprints.

SUMMARY:
The purpose of this study is to investigate the acute effects of different intensities (i.e., 50, 75, and 100% of maximal anaerobic power) of 4-s sprint interval exercise on physiological responses. Secondly, it will determine the relationship between intensity and recovery duration (i.e., 15, 30, or 45-s) that will stimulate the cardiovascular and metabolic systems.

DETAILED DESCRIPTION:
Background Short sprint interval training (sSIT) is typically performed at maximal intensity, generating power far above what is needed to reach peak oxygen consumption (VO₂peak). However, the physiological effects of submaximal sprint intensities and different recovery periods are not well understood.

Study Aim This study examined how power output and oxygen consumption (VO₂) respond to repeated 4-second sprints at 50%, 75%, and 100% of maximal power (Pmax) with rest periods of 15, 30, or 45 seconds.

Methods Eleven recreationally active participants completed nine trials, each consisting of thirty 4-second cycling sprints under different intensity and recovery conditions.

ELIGIBILITY:
Inclusion Criteria:

* Young (18-30),
* Healthy,
* Recreationally active, but untrained (not meeting ACSM's recommendations of 150 min/week of moderate-vigorous aerobic exercise)

Exclusion Criteria:

* Cardiovascular disease
* Smoking
* Subjects who were exercising regularly (>75 min/week) were excluded.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Cardiovascular changes | From enrollment (Day 1) to the end of treatment (9 trials) (Day 11), through study completion, an average of 5 weeks.
  The %VO2peak associated with repeated submaximal power sprints (%Pmax), particularly when paired with varying rest periods, remains unknown. The aim of this study was to systematically investigate the cardiovascular changes for better exercise programming, measured in mL/min/kg.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Laboratory, Department of Kinesiology and Health Education, the University of Texas at Austin, Austin, Texas, United States